CLINICAL TRIAL: NCT06851234
Title: Fluid Dynamics of Concussion in Mixed Martial Arts in a Pilot Randomized Controlled Trial of Osteopathic Manipulative Medicine
Brief Title: Osteopathic Manipulative Treatment RCT and Computational Modeling for Head Injuries in Mixed Martial Artists
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHS2024 135; 24007886 (Other Grant/Funding Number: American Osteopathic Association)
Record Dates: First submitted 2025-01-17; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Head Injury Trauma
Keywords: osteopathic manipulative treatment; concussion; mixed martial arts; head injury
MeSH Terms: conditions — Brain Concussion; Craniocerebral Trauma | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The pre-fight outcome measures, computational modeling of any head injury during the fight, and the post-fight outcome measures will be done on all research participants. If the participant did sustain a head injury or concussion, then, they would be randomly put in the OMM treatment or Sham treatment groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding: The investigators measuring cognitive neuropsychology and computational modeling will be blinded to grouping, and the investigators performing the OSE will be blinded to each others' diagnoses as well as the other outcome measures. If there are any concerns for health identified on cognitive neuropsychology testing, Dr. Amber Sousa, Ph.D is a clinical neuropsychologist who can direct participants for appropriate care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathic manipulative medicine (OMM) (Experimental): Intervention Goals: The varied vectors of head injuries potentially leading to concussion necessitate the initial (Part A) techniques to be individualized to the participant and their OSE. Part B is required techniques to optimize lymphatic and/or glymphatic circulation as outlined below. All investigators (JDM, RAS, PK) who perform OMM will meet to discuss treatment approaches to best achieve consistency.
  1. Cranial 15 min. Part A: treatment of any new somatic dysfunctions and cranial lifts for suture compressions.
     Part B: Thoracic outlet release, OA decompression, V-Spread, Venous sinus drainage, cranial-OMM for strain patterns, facial effleurage, and Cranial treatments will end with a CV4.
  2. Spine 5 min. Use of appropriate techniques for the dysfunctions, such as Balanced ligamentous tension (BLT), muscle energy techniques, facilitated positional release, articulatory techniques (ART), high-velocity low-amplitude, and counterstrain.
  3. Rib Cage 5 min.
  4. Sacrum/Pelvis 5 min.
  Interventions: Procedure: osteopathic manipulative medicine
- Control (Sham Comparator): Sham-Light-Touch Control 30 minute sessions
  Interventions: Procedure: The sham light touch will be performed by an investigator not trained in bodywork or a first--year osteopathic medical student.

INTERVENTIONS:
Procedure: osteopathic manipulative medicine — OMM
  Arms: Osteopathic manipulative medicine (OMM)
Procedure: The sham light touch will be performed by an investigator not trained in bodywork or a first--year osteopathic medical student. — Participants will lay supine on an OMM table. After the OSE, the investigator will place their hands flat in light contact with the participants' parietal bone regions, then the shoulders, then the sides of the lower ribs, and finally over the trochanters.
  Arms: Control

SUMMARY:
The purpose is to test how osteopathic medicine (OMM) improves recovery after a hit to the head during Mixed Martials Arts (MMA). The small changes in the bone, joints, and fluids during head injuries may lead to traumatic brain injury (TBI). The OMM is adjusting the body with the doctors' hands. The goal is to restore alignment and release tension. The head is treated with the doctors' hands placed gently on the head or face. It was previously found to improve symptoms and recovery of memory after head injuries in college athletes. There haven't been clinical trials of this procedure in MMA fighters. Yet, they often get injuries to the part of the brain that releases hormones. Referrals for tests for the hormones are available. Individuals who participate in MMA fighting or sparring matches may join this study. Those who don't get hit in the head or a concussion will contribute to our understanding the osteopathic structural physical exam and fluid dynamics of the head in relation to brain function tests. Those who get hit in the head may be put in the treatment procedure or sham-placebo group. Participants will not be told which group they are in. We anticipate that 100 individuals of any gender will enroll in this study at NYIT Academic Health Care Center (AHCC). To be in this study, the participant must:

Part 1 - Before the fight:

1. Plan to participate in an MMA fight or sparring match,
2. 18 to 50 years of age,
3. Be able to do online cognitive neuropsychology tests for memory, reaction time, and symptoms.

Part-2-After the fight:

(1) Have been hit in the head, or had a head injury, during a fight

The participant cannot be in this study if they have:

Part 1- Before the fight:

1. a current or previous spinal cord injury,
2. a traumatic brain injury within the past six months,
3. inability to tolerate the sports physical,
4. a diagnosis of brain degeneration,
5. low hormones levels from the brain,
6. Pregnancy Participants won't get referred for hormone testing if they don't have any clinical signs of this injury. They also won't get referred for it if they've had heart disease, disease of the blood vessels in their brain, or seizures.

Participants cannot be in Part-2-After the fight if they:

1. cannot tolerate OMM (For example, you have a skull fracture, cervical spine fracture, bleeding or increased pressure in the head, tearing of tissues in the neck, space-occupying lesion, or stroke).
2. were knocked out for more than 2 minutes, had seizures, persistent vomiting, or paralysis when your head was hit.

Participation involves 2 or 4 visits, which will take place over one week.

* The first visit takes 30 mins. in-person and 70 mins. of online testing from home.
* The second visit takes 30-60 mins. in-person and 70 mins. of online testing from home.
* The third & fourth visits will each be 30 mins. in-person and 70 mins. online testing from home.

If participants agree to be in this study, they will be asked to do the following:

Visit #1: Before the Fight

* Get screened and review the consent form
* Take the neuropsychology tests (ImPACT and Inquisit Web) online from home
* Get a non-invasive sports physical exam of head, neck, back, arms, and legs.
* Urine sample for the hormone from the brain called oxytocin (optional)
* Have blood sugar checked by a lancet after pricking the finger (optional) Fight video: The study-doctors will record the participants' fights to make a computational model of the head.

Visit 2: After the Fight

* Get a sports physical of head, neck, back, arms, and legs.
* IF the participant was hit in the head, the study-doctors or participants private doctor will examine them.
* Take the ImPACT and Inquisit Web tests online from home
* If the participant had an injury to their brain, they may get the OMM procedure or sham placebo-control (non-therapeutic light touch).
* Urine sample for the hormone from the brain called oxytocin (optional)
* Have your blood sugar checked by a lancet after pricking your finger (optional)
* Referral to your doctor to test the levels of other brain hormone (optional)

Visit 3 & 4:

* Sports physical of head, neck, back, arms, and legs
* Take the ImPACT and Inquisit Web tests online from home
* If you had an injury to your brain, you may get the OMM procedure or sham placebo-control (nontherapeutic light touch). You will not be told which one you are getting.
* Urine sample for oxytocin (optional)
* Have blood sugar checked by a lancet after pricking your finger (optional)
* Referral to test the levels of other brain hormone (optional) Any significant new findings that develop during research that may relate to the participants health or willingness to continue will be provided to them by phone call. The results will help us understand head injuries, how well OMM works to treat them, and may improve future care for fighters.

DETAILED DESCRIPTION:
Investigating the benefits of osteopathic manipulative medicine (OMM) on head injury has the potential to advance the knowledge and application of osteopathy. Traumatic brain injury (TBI) including concussion, or mild traumatic brain injury (mTBI), is an injury resulting from a force directed towards the head that precedes and contributes to new onset symptoms and/or impairments in cognitive neuropsychology without discrete lesions detectable by traditional imaging. Its annual financial burden in the United States (USA) is $1.4-3.8 million, and there are limited treatments. Current practice guidelines (CPG) recommend rest with gradual return-to-play. Mixed martial artists (MMA) often sustain head injuries during fights or sparring matches, and they experience changes in cognitive neuropsychological testing. Faster recovery from symptoms and in visual memory and reaction time were found after OMM in a randomized controlled trial (RCT) in college athletes with acute uncomplicated concussions utilizing the same OMM methods in this proposal for use in MMA. This OMM sequence was previously outlined by the P.I. in 2016. The OMM treatment sequence addresses structural restrictions throughout the whole body, including improving glymphatic and venous circulation of the brain to allow for self-regulation, self-healing, and health maintenance. The purpose of this study is to test if OMM significantly improves symptoms and cognitive recovery after head injury during mixed martial arts (MMA) fights compared to a sham control group. Hypothesis: Participants with concussion during an MMA fight have significantly better recovery in neuropsychological tests and symptoms after receiving three OMM treatments compared to those receiving three Sham-Light touch control sessions over 1-week.

Aim 1: Determine if there is significant improvement in head injury-related impairments on ImPACT and Inquisit Web measures in individuals after three OMM sessions compared to three Sham-Light touch Aim 2: Determine if Pre-fight to Post-fight changes in cranial strain patterns are significantly correlated with ImPACT or Inquisit Web changes in individuals with head injuries during a recorded fight.

Aim 3: Test for significant associations between cranial strain patterns, forces causing injury, neuropsychologicalmeasures, and brain region impacted upon coup-contrecoup of the brain. Eligible, consented participants of any gender will be recruited for Part-1 of this study, which is an observation study of head injury dynamics and epidemiology; it doesn't include an intervention. Participants with concussion symptoms due to head injury during MMA fights within the preceding three (3) days will continue to Part-2-Interventions and be randomized into OMM or Sham-Light-touch control groups. Pre- to Post-Injury changes on ImPACT, Inquisit Web, and cranial strain patterns will be tested for significant correlations with the brain area impacted upon contrecoup according to the computational model. Post-Injury changes and Post-interventions tests will be compared utilizing a generalized linear model (GLM) by NYITCOM biostatistician.

Main study outcome measures:

1. The detailed physical examination for performing OMM is referred to as the osteopathic structural exam (OSE) for somatic dysfunctions, and OMM involves non-invasive manual treatments of the somatic dysfunctions to improve physiologic function. The OSE can reveal potential cranial somatic dysfunctions after concussion. Examining the cranium for somatic dysfunctions involves assessing sphenobasilar synchondrosis (SBS) biomechanics. The physiologic SBS somatic dysfunctions, sidebending rotation (SBR) or torsion patterns, are common and can happen organically. Sidebending of SBS somatic dysfunctions occurs around two vertical axes with rotation around an anteroposterior axis. Torsion occurs around an anteroposterior axis as well.

   Conversely, nonphysiologic SBS somatic dysfunctions include vertical or lateral shears and/or compression patterns, which are less common. Lateral shears occur around two vertical axes, whereas vertical shears occur around two transverse axes. Research suggests that nonphysiologic somatic dysfunctions typically result from physical trauma and rarely resolve on their own.
2. Computational CSF dynamics
3. ImPACT : The computerized ImPACT measures visual memory (Visual), verbal memory (Verbal), visual-motor processing speed (PS), reaction time (RT), impulse control (IC), and patient-rating of symptom severity (SS). It's a well-established, validated tool widely utilized for measuring cognitive function following concussion injury. The ImPACT had 81.9% sensitivity and 89.4% specificity in detecting concussion-related new onset impairments (NOI) when administered during the pre-participation sports physical to establish Baseline, and, again, after sustaining a concussion (Post-Injury), compared to normalized, validated age-gender-matched demographic data. The demographic data section of ImPACT includes relevant sport, medical, and concussion history information.

   The Inquisit Web (Millisecond Software LLC, Seattle, WA, USA) is another computer-based platform that allows for the administration of neuropsychological tests specifically for acute changes in information processing speed, inhibition, and visual and verbal learning memory tasks with a delayed memory recall.
4. Oxytocin ELISA

Inclusion criteria:

Part 1-head injury dynamics:

* (1) individuals participating in MMA fights or sparring matches,
* (2) 18 to 50 years of age,
* (3) able to complete online cognitive neuropsychology tests.

Part-2-Intervention:

- (1) having a witnessed closed head injury during a fight exclusion criteria.

Part 1-head injury dynamics:

* (1) having a current or previous spinal cord injury,
* (2) head injury within past six months,
* (3) being unable to complete the assessment,
* (4) been diagnosed with underlying neurodegenerative condition,
* (5) pre-existing hypopituitary function,
* (6) Pregnancy.

Part-2-Intervention:

* (1) has absolute contraindications to OMM (e.g. skull fracture, cervical spine fracture, signs of intracranial bleeding or increased intracranial pressure, cervical dissection, space occupying lesion in the cranium, or stroke),
* (2) suffered a witnessed loss of consciousness (LOC) for greater than 2 minutes, seizures, intractable vomiting or paralysis at the time of the head injury.

Participants won't be referred to their private doctors for additional pituitary hormone testing unless there are clinical signs. The optional referral for growth hormone and other pituitary testing by glucagon stimulation Test at Quest labs will be contraindicated if there is risk of and/or a history of (1) cardiovascular (heart) disease, (2) disease of the blood vessel in your brain, or (3) seizures.

The investigators measuring cognitive neuropsychology and computational modeling will be blinded to grouping, and the investigators performing the OSE will be blinded to each others' diagnoses as well as the other outcome measures. If there are any concerns for health identified on cognitive neuropsychology testing, Dr. Amber Sousa, Ph.D is a clinical neuropsychologist who can direct participants for appropriate care.

Eligible, consented participants of any gender will be recruited for Part-1 of this study, which is an observation study of head injury dynamics and epidemiology; it doesn't include an intervention. Participants with concussion symptoms due to head injury during MMA fights within the preceding three (3) days will continue to Part-2-Interventions and be randomized into OMM or Sham-Light-touch control groups. Pre- to Post-Injury changes on ImPACT, Inquisit Web, and cranial strain patterns will be tested for significant correlations with the brain area impacted upon contrecoup according to the computational model. Post-Injury changes and Post-interventions tests will be compared utilizing a generalized linear model (GLM) by NYITCOM biostatistician.

Computerized cognitive neuropsychological tests:

The ImPACT is a widely used test that will be administered to athletes 12 years of age or older before sports to establish a baseline of cognitive function, and administered again with the suspicion of a brain injury to evaluate differences in cognitive function. ImPACT has been shown to be an effective adjunctive test for evaluation of concussion as part of a comprehensive medical diagnosis involving other testing methods. The positive predictive value (PPV-probability that a concussion is present when the test is positive) is 89.4% and the negative predictive value (NPV-probability that a concussion is not present when the test is negative) is 81.9% (Schatz 2006). ImPACT is a 25-minute online test to be administered through a secure web portal by a licensed healthcare provider. ImPACT will be administered via a link on a computer in a quiet office room according to the ImPACT guidelines, through the P.I.'s login. A new profile will be created for each participant by their study-participant#.

Participants will take a 4 hour break after ImPACT to minimize computer-use stress both pre- and post-fight for more consistent data. If a participant's IC index is elevated on the baseline testing, the participant will be asked to retest, and test-retest reliability computation will be done.

Lower reliability estimates (lower ICCs) were observed in a study utilizing the more stringent validity criteria of IC composites greater than 20 (Resch et al., 2013). The main aim of the IC index is Response Inhibition or Delay (Schatz 2006), however, the IC has been reported to be high at baseline due to a several factors. These include 'sandbagging' (purposing getting lower baseline score to avoid seeming like having a concussion Post-injury), Left-Right confusion, trouble with sleep, and oculomotor disorders (IC>20) (Brett et al 2016, Schatz 2006, Mancini 2022). Re-testing for reliability has been found useful in previous research publications.

Then, participants will complete cognitive testing via the Inquisit Web (Millisecond Software LLC, Seattle, WA, USA) platform. This platform is a computer-based platform that allows for the administration of neuropsychological tests specifically for acute changes in information processing speed, inhibition, and word learning tasks with a delayed-recall. Measures from the platform that will be included are the Paced Auditory Serial Addition Test (PASAT) (8 min.), Continuous Performance test (20 min.), and Rey Visual Design Learning Test (15 min.). Participants will take a 5 min. break between tests. The PASAT is a measure of information processing speed in which participants listen to a string of digits and mentally sum the last two. The Continuous Performance Test is a test of sustained and selective attention. The Verbal Selective Reminding test is a 12- list word learning task with a delay recall condition. The Rey Visual Design Learning Test assesses visual memory. The total testing time is expected to be 69 minutes with break-time.

Inquisit Millisecond Measures Paced Auditory Serial Addition Test (PASAT) - 8 min. script implements a computerized version of the Paced Auditory Serial Addition Test (PASAT), a measure of information processing rate. Participants hear a sequence of single digit numbers (1-9) presented at a constant speed and are asked to mentally sum the last 2 digits (NOT a running total). Participants then select the current sum from a circle of numbers 1-18 (= nonverbal response) The implemented procedure is based on Gronwall, D. 1977.

Continuous Performance Test- 20 min. is for sustained and selective attention. Participants get presented a sequence of letters (one-by-one). Task1: press the Spacebar whenever the letter is an X Task2: press the Spacebar whenever the letter is an X that follows an A. Rosvold, et al. 1956. Rey Visual Design Learning Test- 15 min. (RVDLT) is an assessment tool for immediate/delayed and recognition memory for non-verbal items. Participants are presented 15 simple figures. Each figure is presented for 2s (default). Afterwards recall (immediate/delayed) and recognition tests are given. The implemented procedure is based on P. Wilhelm 2004.

Inquisit Tests licensed:

Verbal Selective Reminding Task- 20 min. is a list learning and free verbal recall test that allows the simultaneous analysis of long term and short-term storage. Participants see a list of 12 words, presented to them one by one, and have to recall as many words as they can by typing all words into the keyboard. For those items that were not recalled during the current trial, the words are repeated and participants are again asked to recall as many of the original list words as they can. This procedure is repeated for 12 trials (Buschke, H. 1973).

Online Tests from home Per Visit Time ImPACT 26 minutes BREAK if needed Paced Auditory Serial Addition Test (PASAT) 8 minutes BREAK if needed Continuous Performance test 20 minutes BREAK if needed Rey Visual Design Learning Test 15 minutes Total online test time 69 Total break time variable

Video-recording of fights:

The tournaments will be video-recorded by the investigators for later computational modeling of head injury for the coup-contrecoup brain regions. The videos will be confidential, only viewable by the investigators. Two tripods to maintain steady camera angles will be used, in addition to a third handheld camera to catch other views. The location of the cameras on tripods may depend on facilities and safety. The investigators will be far enough away from the fight ring to avoid accidental injury (>5 ft.) Computation of the model takes 1-7 days depending on how complicated the injury vectors are.

Participants with concussion due to head injury during the MMA matches within the preceding 2 days will be interviewed and evaluated by the physician-investigators (Jayme Mancini, DO, Ph.D, P. Kooyman, DO, or Reem Abu-Sbaih, DO) to confirm the diagnosis. The MACE will be used if the evaluation for concussion diagnosis is unclear. Any individuals having signs of concussion complications requiring emergency care will be directed to emergency services. Participants will be encouraged to also see their primary care or sports medicine providers if they haven't already seen them or the emergency department.

All care that participants receive other than in the proposed study will be documented and tested statistically for interaction with the results. The CPG of rest from activity will be recommended for those concussed.

Participants may opt in for a urine sample collection in urine cups during the visits to be preserved and frozen for later oxytocin concentration analysis by Satoru Kobayashi, Ph.D.

Urine sample collection will also be done directly after the two intervention visits. They'll be stored in the -80 freezer in Riland Building room 23. In this proposed study, the post-fight assessment of head injury will include muscle testing for pituitary function. If there are clinical signs of pituitary injury, the investigators will refer participants to their private doctor for diagnosis of head trauma and recommendation of the glucagon stimulation test. For those individuals having suspicion of hypopituitary function or having new Post-Injury nonphysiologic SBS dysfunctions. The investigators will refer participants for a Glucagon Stimulation Test at Quest or other labs.

Osteopathic Physical Exam & OMM The OMM Group participants will receive a 30-minute OSE and treatment session detailed below. Two licensed osteopathic physicians board certified in neuromusculoskeletal medicine will perform an OSE of the head for interrater reliability, and one physician will perform the 30 minute treatment session. Then, participants will follow up for a second treatment 48-72 hours post-1st - visit. Sham control group participants will receive a 30-minute sham light touch session. Then, participants will follow up for a second sham session 48-72 hours post-1st-visit. The OMM will be performed by the physician-investigators (JM, RAS, PK) in an outpatient room at site NYIT AHCC.

Osteopathic Physical Exam & OMM

The OMM Group participants will receive a 30-minute OSE and treatment session detailed below. Two licensed osteopathic physicians board certified in neuromusculoskeletal medicine will perform an OSE of the head for interrater reliability, and one physician will perform the 30 minute treatment session. Then, participants will follow up for a second treatment 48-72 hours post-1st - visit. Sham control group participants will receive a 30-minute sham light touch session. Then, participants will follow up for a second sham session 48-72 hours post-1st-visit. The OMM will be performed by the physician-investigators (JM, RAS, PK) in an outpatient room at site NYIT AHCC. OSE and documentation for severe or key somatic dysfunctions will include:

1. Cranial & Face - Assess for somatic dysfunctions of SBS (SBR, torsion, lateral, vertical), palatine, zygoma, and other strain patterns, Occipitoatlantal (OA) joint, compressed sutures, Cranial rhythmic impulse (CRI), osteopathy in the cranial field, and intraosseous strains. The palatine bones act as tensioners, while the zygoma bones function as dampeners to the CRI.
2. Spine - cervical, thoracic, and lumbar
3. Rib Cage - ribs, thoracic outlet, sternal-clavicle dysfunction, thoracic diaphragm
4. Sacrum and Pelvis

Testing cranial strain patterns:

The pre-fight osteopathic physical exam (OSE) of the head will be performed by two boardcertified, licensed physicians using their hands for diagnosis of somatic dysfunctions of sphenobasilar synchondrosis (SBS) (1. compressed, 2. SBR, 3. torsion, 4. lateral, 5. Vertical, 6. Physiologic), palatine and zygoma (1. inhalation or 2. Exhalation), other severe strain patterns, condylar compression, occipitoatlantal (OA) joint (flexion or extension), and severely compressed sutures as well as cranial rhythmic impulse (CRI), osteopathy in the cranial field, and intraosseous strains. The vault or the Becker-holds will be used to palpate the head. Participants sustaining a concussion from a head injury during the fight will be randomly assigned into groups receiving two OMM treatments or two sham-light-touch control sessions.

OMM Group Intervention Goals: The varied vectors of head injuries potentially leading to concussion necessitate the initial (Part A) of treatment techniques to be individualized to the participant and their OSE. Then, (Part B) there are several required techniques to optimize lymphatic and/or glymphatic circulation as outlined below. All the investigators (JDM, RAS, PK) who perform OMM will meet to discuss treatment approaches in order to best achieve consistency.

1. Cranial 15 min. - Part A: treatment of any new somatic dysfunctions and cranial lifts for suture compressions.

   Part B: Thoracic outlet release, OA decompression, V-Spread, Venous sinus drainage, cranial-OMM for strain patterns, facial effleurage, and Cranial treatments will end with a CV4. (Chapter 18: Osteopathic Cranial Manipulative Medicine. Atlas of Osteopathic Techniques, 3e.). https://meded-lwwhealthlibrarycom
2. Spine 5 min. - Use of appropriate techniques for the dysfunctions, such as Balanced ligamentous tension (BLT), muscle energy techniques, facilitated positional release, articulatory techniques (ART), high-velocity low-amplitude, and counterstrain 3. Rib Cage 5 min. - Thoracic outlet release (TOR) will be performed first. Any additional rib cage dysfunctions can be addressed with rib raising, ART, or any other standard OMM.

4. Sacrum/Pelvis 5 min. - Address dysfunction with appropriate standard OMM. Sham-Light-Touch Control 30 minute sessions: The sham light touch will be performed by an investigator not trained in bodywork or a first- or second-year osteopathic medical student. Participants will lay supine on an OMM table. After the OSE, the investigator will place their hands flat in light contact with the participants' parietal bone regions, then the shoulders, then the sides of the lower ribs, and finally over the trochanters. Treatment and Sham sessions will be performed in the patient care rooms at NYIT AHCC.

Coup-contrecoup Neuroanatomy Determined by Individual Participant Fluid-Structure Interaction Analyses of Cerebrospinal Fluid Interacting with Brain using Computational Simulations:

1. Material and Methods The type of studies conducted using this method falls under the definition of a single case study where one type of patient specific geometry is considered in combination with one type of boundary and initial conditions. The geometry, computational method, and boundary conditions used are introduced as follows.

1.1. Geometrical Model The head model used consists of numerous parts, namely, the cerebrum, cerebellum, brainstem, pituitary, skull, and the fluid particles prescribed to fill the space between all the brain parts and the skull (i.e., subarachnoid space). The helmet placed on the skull has two layers, namely, thicker deformable padding and a thinner hard-shell cover. The foam padding is tightly fitting on the skull with no skull/ helmet gaps.

1.1. Computational Methods Smoothed-Particle Hydrodynamics (SPH) is a computational meshfree Lagrangian method developed in 1977, initially for astrophysical problems. Since then, it has been used for simulating the mechanics of continuum media, such as solid mechanics and fluid flows. It has been used in many fields outside astrophysics, e.g. ballistics, volcanology, and oceanography. Increasingly, it is being adopted by many with an interest in biomedical engineering. Fluid motion and boundary interaction calculations were subsequently solved with the IMPETUS Afea Solver using SPH for the fluid domain and the high-order finite element method for the solid domain. Amore detailed description including the formulation used can be found in our prior publications. The model and methods used were previously validated against cadaveric experimental data.

1.2. Boundary Conditions Boundary conditions are applied to the aforementioned model to copy real-life accident/contact scenarios in order to study the consequent interaction between the brain and the cerebrospinal fluid surrounding it. To summarize, the acceleration data extracted from the recordings are used in the IMPETUS Afea Solver to create simulations using the aforementioned models during the ischarge. The SPH is used for the calculations. It is a computational meshfree Lagrangian method, initially developed for astrophysical problems. Since then, it has been used for simulating the mechanics of continuum media, such as solid mechanics and fluid flows. It has been used in many fields outside of astrophysics, e.g., ballistics, volcanology, and oceanography. Increasingly, it is being adopted by many with interest in biomedical engineering The combination of SPH methods used to simulate the fluid domain flow with a high-order finite element method used to simulate the solid domain deformations is ideal for simulating fluid-structure interactions (FSI), especially when complex geometries are included. SPH methods provide numerical stability because the contact between the solid and fluid domains is easily treated numerically. Moreover, SPH is highly parallelizable. That being the case, it is possible to run FSI simulations that are numerically stable, precise, and parallelized on a standard GPU workstation.

We expect that the prospective results from this study will demonstrate the ability to compute the affected brain region that significantly correlates with cranial somatic dysfunctions as well as the cognitive neuropsychology tests. This would also provide insight into the mechanisms underlying concussion and OMM.

Baseline, Post-injury, and Post-interventions measures will be tested statistically by NYITCOM biostatistician. Qualitative measures of past medical history and history of present illness will be evaluated for potential differences in subtypes and confounding variables. Kappa statistics to compare Pre- and Post-Fight inter-examiner concordance of OSE will be computed for interrater reliability. Correlations between variables, covariates, confounding variables will be tested for significance (p<.05). The Spearman rank-order correlation coefficient (rs (or ρ, pronounced rho) is a nonparametric measure of the strength and direction of association that exists between two variables measured on either ordinal variables or for continuous data that has failed the assumptions necessary for conducting the Pearson's product-moment correlation. Spearman's correlations among the measures of the cranial OSE, neuroanatomy injured by contrecoup brain motion based on computational model, and neuropsychological tests will be calculated. Rho (Strength of r: +1 -1 Perfect; +0.9 -0.7 Strong; +0.6-0.4 Moderate; +0.3-0.1 Weak; 0 0 Zero/ None).

ImPACT indices will be statistically tested according to the validated age-gender groups. In previous studies, Control group memory composite scores did not increase with multiple testing opportunities, indicating that the ImPACT memory composite was not hindered by a practice effect (multiple times taking exam) (Schatz 2006). To determine concussion injury effects, differences in ImPACT indices and Inquisit Millisecond Web from Pre-fight to Post-fight will be compared by two-tailed, repeated- measures analysis of variance (ANOVA) with appropriate posthoc test, and symptom scores will be compared for participants with head trauma during the fight versus those without using the Mann-Whitney U test. Among participants with head trauma, those with versus without LOC will be compared similarly. Intraclass correlation coefficient (ICC) will examine agreement between Pre-fight and Post-fight scores among participants without head trauma. The relationships between pre-intervention measures will be determined using Spearman rank correlations.

The recovery rate between groups will be tested by ANOVA for Baseline, Injury, Post-1-Intervention, and Post-2 Intervention cognitive neuropsychology tests. If there is high attrition for the second visit-intervention, the differences in recovery between the groups will also be tested utilizing generalized estimating equations (GEE) for repeated measures. Additionally, for the nonparametric data, related samples Wilcoxon signed-rank test may be utilized to test the null hypothesis that the median of the differences between the Injury and Post-2 Intervention within-group outcome equals 0. Potential covariates will be tested using Fisher's exact or chi-square test for categorical variables and t-test or ANOVA. Logistic regression will be used to examine baseline predictors of outcome. Predictors could include baseline cognition, pituitary function, baseline symptoms.

The results will increase the understanding of which regions of the head to target treatments, and they would support the use of OMM in the treatment of concussion in MMA while explaining some of the underlying mechanisms of cranial OMM.

ELIGIBILITY:
Inclusion Criteria:

* Part 1-head injury dynamics:

  1. individuals participating in MMA fights or sparring matches,
  2. 18 to 50 years of age,
  3. able to complete online cognitive neuropsychology tests.

     Part-2-Intervention:

  <!-- -->

  1. having a witnessed closed head injury during a fight

     Exclusion Criteria:
* Part 1-head injury dynamics:

  1. having a current or previous spinal cord injury,
  2. head injury within past six months,
  3. being unable to complete the assessment,
  4. been diagnosed with underlying neurodegenerative condition,
  5. pre-existing hypopituitary function,
  6. Pregnancy.

Part-2-Intervention:

1. has absolute contraindications to OMM (e.g. skull fracture, cervical spine fracture, signs of intracranial bleeding or increased intracranial pressure, cervical dissection, space occupying lesion in the cranium, or stroke),
2. suffered a witnessed loss of consciousness (LOC) for greater than 2 minutes, seizures, intractable vomiting or paralysis at the time of the head injury, Participants won't be referred to their private doctors for additional pituitary hormone testing unless there are clinical signs. The optional referral for growth hormone and other pituitary testing by glucagon stimulation Test at Quest labs will be contraindicated if there is risk of and/or a history of (1) cardiovascular (heart) disease, (2) disease of the blood vessel in your brain, or (3) seizures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Osteopathic structural exam | 1 week
  Osteopathic structural exam is a detailed physical exam of the biophysical characteristics such as biomechanical alignment. Testing will be done pre-fight, post-fight, and after the two follow up visits.

SECONDARY OUTCOMES:
ImPACT and Inquisit Web cognitive neuropsychology tests | 1 year
  ImPACT and/or Inquisit Web neuropsychological testing. Testing will be done pre-fight, post-fight, and after the two follow up visits.

OTHER OUTCOMES:
Brain region found at the point of cerebrospinal fluid flux during contrecoup of brain during head injury | 3 days
  The brain region likely affected by contrecoup determined by Individual Participant Fluid-Structure Interaction Analyses of Cerebrospinal Fluid Interacting with the brain using computational simulation models. The fight will be video-recorded, and this outcome measure is based on the videos of any head injury during the fight.

CONTACTS AND LOCATIONS:
Overall Officials: Jayme Mancini, D.O., Ph.D, FAWM, Principal Investigator — New York Institute of Technology College of Osteopathic Medicine, Academic Health Care Center, Riland Building; Amber Sousa, Ph.D, Study Director — New York Institute of Technology College of Osteopathic Medicine; Reem Abu-Sbaih, D.O., Study Chair — New York Institute of Technology College of Osteopathic Medicine
Locations (1):
- Academic Health Care Center of NYIT College of Osteopathic Medicine, Greenvale, New York, United States